CLINICAL TRIAL: NCT01379937
Title: Safety and Immunogenicity Study of a Prime-boost Schedule of GSK Biologicals' Influenza Vaccine GSK1562902A in Children Aged 3 to 17 Years
Brief Title: A Study to Evaluate the Safety and Immunogenicity of a Prime-boost Schedule of GSK Biologicals' Influenza Vaccine in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 115115
Record Dates: First submitted 2011-06-17; First posted 2011-06-23 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2016-08

CONDITIONS: Influenza
Keywords: influenza; H5N1; vaccine; children
MeSH Terms: conditions — Influenza, Human | interventions — Hepatitis A Vaccines

ARMS (4):
- GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group (Experimental): Subjects in this group received 2 primary vaccination doses of Influenza vaccine GSK1562902A Formulation 1, a booster vaccination dose of Influenza vaccine GSK1562902A Formulation 2 and 1 dose of Havrix™ or Havrix™ Junior vaccine, administered intramuscularly in the deltoid region.
  Interventions: Biological: Influenza vaccine GSK1562902A Formulation 1; Biological: Influenza vaccine GSK1562902A Formulation 2; Biological: Havrix™; Biological: Havrix™ Junior
- GSK1562902A Formulation 1 - Havrix / Havrix Jr Group (Experimental): Subjects in this group received 2 primary vaccination doses of Influenza vaccine GSK1562902A Formulation 1 and 2 doses of Havrix™ or Havrix™ Junior vaccine, administered intramuscularly in the deltoid region.
  Interventions: Biological: Influenza vaccine GSK1562902A Formulation 1; Biological: Havrix™; Biological: Havrix™ Junior
- GSK1562902A Formulation 2 - Havrix / Havrix Jr Group (Active Comparator): Subjects in this group received 1 dose of Influenza vaccine GSK1562902A Formulation 2 and 2 doses of Havrix™ or Havrix™ Junior vaccine, administered intramuscularly in the deltoid region.
  Interventions: Biological: Influenza vaccine GSK1562902A Formulation 2; Biological: Havrix™; Biological: Havrix™ Junior
- Havrix / Havrix Jr Group (Active Comparator): Subjects in this group received 2 doses of Havrix™ or Havrix™ Junior vaccine, administered intramuscularly in the deltoid region.
  Interventions: Biological: Havrix™; Biological: Havrix™ Junior

INTERVENTIONS:
Biological: Influenza vaccine GSK1562902A Formulation 1 — Intramuscular injection, two doses each in GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group and GSK1562902A Formulation 1 - Havrix / Havrix Jr Group
  Arms: GSK1562902A Formulation 1 - Havrix / Havrix Jr Group; GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group
Biological: Influenza vaccine GSK1562902A Formulation 2 — Intramuscular injection, one dose each in GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group and GSK1562902A Formulation 2 - Havrix / Havrix Jr Group
  Arms: GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group; GSK1562902A Formulation 2 - Havrix / Havrix Jr Group
Biological: Havrix™ — Intramuscular injection, one dose in GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group and two doses each in GSK1562902A Formulation 1 - Havrix / Havrix Jr Group, GSK1562902A Formulation 2 - Havrix / Havrix Jr Group and Havrix / Havrix Jr Group
Biological: Havrix™ Junior — Intramuscular injection, one dose in GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group and two doses each in GSK1562902A Formulation 1 - Havrix / Havrix Jr Group,GSK1562902A Formulation 2 - Havrix / Havrix Jr Group and Havrix / Havrix Jr Group

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity of a prime-boost schedule of GSK Biologicals' influenza vaccine in children aged 3 to 17 years.

DETAILED DESCRIPTION:
In this study Influenza vaccine GSK1562902A is the primary study vaccine and Havrix™ will be administered as the active comparator and not co-administered along with the study vaccine.Therefore, there exist no relation between the vaccines administered in this study. As the study will be carried out in Philippines, Havrix™ vaccine will be used as an active comparator instead of saline placebo to offer an advantage to the subjects.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy ALL the following criteria at study entry:

* Subjects for whom the investigator believes that the parent(s)/Legally Acceptable Representative(s) [LAR(s)] can and will comply with the requirements of the protocol .
* A male or female child 3 to 17 years of age inclusive, at the time of the first vaccination.
* Written informed consent obtained from the subject's parent or guardian. Assent obtained from the subject when applicable.
* Good general health as established by medical history and clinical examination before entering into the study.
* Comprehension by the subject's parent or guardian of the study requirements, ability to comprehend and comply with procedures for collection of short- and long-term safety data, expressed availability for the required study period, and ability and willingness to attend scheduled visits.
* Parent/LAR with access to a consistent means of telephone contact, land line or mobile, but NOT a pay phone or other multiple-user device (i.e., a common-use phone serving multiple rooms or apartments).
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

The following criteria should be checked at the time of study entry. If ANY exclusion criterion applies, the subject must not be included in the study:

* Child in care
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of the study vaccine or planned use during the study period.
* Planned administration of any vaccine 30 days prior and 21 days after any study vaccine administration.
* Active participation in other clinical trials.
* Receipt of systemic glucocorticoids within 1 month prior to study enrollment, or any other cytotoxic or immunosuppressive drug within 6 months of study enrollment. Topical, intra-articular or inhaled glucocorticoids are allowed.
* Acute disease and/or fever at the time of enrolment:
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination (no laboratory testing required).
* Acute or chronic, clinically-significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by medical history and physical examination.
* An acute evolving neurological disorder or history of Guillain-Barré syndrome within 6 weeks of receipt of seasonal influenza vaccine.
* Receipt of any immunoglobulins and/or any blood products within 9 months of study enrolment or planned administration of any of these products during the study period.
* Any known or suspected allergy to any constituent of influenza vaccines ; a history of anaphylactic-type reaction to vaccine components or a history of severe adverse reaction to a previous influenza vaccine.
* History of seizures or progressive neurological disease.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Diagnosed with cancer or any chronic severe disease.
* Previous administration of any H5N1 vaccine.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 520 (Actual)
Dates: Start 2011-07-28; Primary Completion 2012-08-02 (Actual); Study Completion 2012-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Philippines (2):
  - GSK Investigational Site, Alabang, Muntinlupa
  - GSK Investigational Site, Quezon City

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Izurieta P, Uy-Aragon MJ, Drame M, Vaughn DW. Assessment of Prime-boost Vaccination Using an AS03B-adjuvanted Influenza A (H5N1) Vaccine: A Randomized Trial in Children of Three to Less Than Eighteen Years of Age. Pediatr Infect Dis J. 2016 Feb;35(2):e35-47. doi: 10.1097/INF.0000000000000968. PMID 26551446
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 115115 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115115 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115115 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115115 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115115 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115115 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was of an overall duration 364 days for all subjects.
Period: Overall Study
Arm/Group | GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group | GSK1562902A Formulation 1 - Havrix / Havrix Jr Group | GSK1562902A Formulation 2 - Havrix / Havrix Jr Group | Havrix / Havrix Jr Group
Started | 156 | 156 | 104 | 104
Completed | 155 | 153 | 102 | 103
Not Completed | 1 | 3 | 2 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Consent withdrawal | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group | GSK1562902A Formulation 1 - Havrix / Havrix Jr Group | GSK1562902A Formulation 2 - Havrix / Havrix Jr Group | Havrix / Havrix Jr Group | Total
Number analyzed (Participants) | 156 | 156 | 104 | 104 | 520
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.70 (4.26) | 9.40 (3.88) | 9.3 (3.87) | 9.6 (4.23) | 9.51 (4.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 81 | 52 | 52 | 266
  Male | 75 | 75 | 52 | 52 | 254

OUTCOME MEASURES:

1. Primary Outcome: Haemagglutination Inhibition (HI) Antibody Titers for the A/Turkey/Turkey/01/2005 (H5N1) Vaccine Strain.
Description: Antibody titers were expressed as Geometric mean titers (GMTs). The H5N1 vaccine strain included A/Turkey/Turkey/01/2005 antigen. The A/Turkey/Turkey/01/2005 (A/TURK) vaccine strain was administered to groups receiving the adjuvanted Influenza vaccine GSK1562902A. This outcome concerns solely subjects in the GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group and GSK1562902A Formulation 2 - Havrix / Havrix Jr Group as required by the protocol.
Time Frame: At Day 192.
Population: The analysis was based on the ATP cohort for immunogenicity, which included all evaluable subjects (i.e., those meeting all eligibility criteria, complying with the procedures and intervals defined in the protocol, with no elimination criteria during the study) and for whom assay results were available for antibodies against the study vaccine.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group | GSK1562902A Formulation 2 - Havrix / Havrix Jr Group
Number analyzed (Participants) | 127 | 84
Titer | 737.6 [646.8 to 841.1] | 24.7 [19.7 to 31.0]

2. Primary Outcome: Number of Subjects With Any Medically Attended Adverse Events (MAEs)
Description: Any = occurrence of the symptom regardless of intensity grade. This outcome concerns solely subjects in the GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group and GSK1562902A Formulation 2 - Havrix / Havrix Jr Group as required by the protocol.
Time Frame: From Day 0 to Day 182
Population: The analysis was based on the Total vaccinated Cohort, which included all subjects with at least 1 vaccine administration documented.
Measure: Number; unit: Subjects
Groups:
- GSK1562902A Formulation 1 & 2 - Havrix/Havrix Jr Pooled Group: Pooled group of subjects who received 2 primary vaccination doses of Influenza vaccine GSK1562902A Formulation 1, no or 1 booster dose of vaccination dose of Influenza vaccine GSK1562902A Formulation 2 and 1 or 2 doses of Havrix™ or Havrix™ Junior vaccine, administered intramuscularly in the deltoid region.
- GSK1562902A Formulation 2 - Havrix/Havrix Jr Pooled Group: Pooled group of subjects who received no or 1 dose of Influenza vaccine GSK1562902A Formulation 2 and 2 doses of Havrix™ or Havrix™ Junior vaccine, administered intramuscularly in the deltoid region.
Arm/Group | GSK1562902A Formulation 1 & 2 - Havrix/Havrix Jr Pooled Group | GSK1562902A Formulation 2 - Havrix/Havrix Jr Pooled Group
Number analyzed (Participants) | 312 | 208
Subjects | 115 | 64

3. Primary Outcome: Number of Subjects With Any Medically Attended Adverse Events (MAEs)
Description: Any = occurrence of the symptom regardless of intensity grade.
Time Frame: From Day 0 to Day 364.
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group | GSK1562902A Formulation 1 - Havrix / Havrix Jr Group | GSK1562902A Formulation 2 - Havrix / Havrix Jr Group | Havrix / Havrix Jr Group
Number analyzed (Participants) | 156 | 156 | 104 | 104
Subjects | 65 | 84 | 41 | 41

4. Secondary Outcome: H5N1 HI Antibody Titres Against the A/Indonesia/5/2005 and A/Turkey/Turkey/01/2005 (H5N1 Virus) Strains
Description: The antibody titres were given as Geometric Mean Titer (GMT). A/Indonesia/5/2005 = A/INDO and A/Turkey/Turkey/01/2005 = A/TURK.
Time Frame: At Days 0, 42, 182, 192, 364
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group | GSK1562902A Formulation 1 - Havrix / Havrix Jr Group | GSK1562902A Formulation 2 - Havrix / Havrix Jr Group | Havrix / Havrix Jr Group
Number analyzed (Participants) | 155 | 152 | 103 | 101
Titer
  A/INDO, Day 0 [N=155,152,103,101] | 5.7 [5.4 to 6.0] | 5.5 [5.2 to 5.8] | 5.4 [5.1 to 5.8] | 5.8 [5.3 to 6.3]
  A/INDO, Day 42 [N=155,152,103,101] | 553.5 [490.9 to 624.1] | 595.0 [522.1 to 678.2] | 5.6 [5.2 to 6.0] | 6.2 [5.6 to 7.0]
  A/INDO, Day 182 [N=155,152,103,101] | 52.2 [47.7 to 57.1] | 54.1 [49.5 to 59.1] | 5.1 [5.0 to 5.2] | 5.6 [5.3 to 6.0]
  A/INDO, Day 192 [N=127,NA,45,NA] | 674.1 [595.0 to 763.8] | NA [NA to NA] — For D192 , antibody titers were tabulated for GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group and GSK1562902A Formulation 2 - Havrix / Havrix Jr Group as required by the protocol. | 7.6 [6.7 to 8.5] | NA [NA to NA] — For D192 , antibody titers were tabulated for GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group and GSK1562902A Formulation 2 - Havrix / Havrix Jr Group as required by the protocol.
  A/INDO, Day 364 [N=151,147,100,NA] | 205.5 [183.3 to 230.4] | 40.4 [36.8 to 44.5] | 8.5 [7.6 to 9.4] | NA [NA to NA] — For D364, antibody titers were tabulated for GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group, GSK1562902A Formulation 1 - Havrix / Havrix Jr Group and GSK1562902A Formulation 2 - Havrix / Havrix Jr Group as required by the protocol.
  A/TURK, Day 0 [N=155,152,103,101] | 7.0 [6.3 to 7.7] | 6.4 [5.9 to 7.0] | 6.1 [5.6 to 6.8] | 7.2 [6.3 to 8.2]
  A/TURK, Day 42 [N=155,152,103,101] | 193.0 [172.1 to 216.5] | 240.3 [188.1 to 240.3] | 6.9 [6.9 to 7.9] | 8.5 [7.2 to 10.0]
  A/TURK, Day 182 [N=127,152,84,101] | 39.6 [35.8 to 43.8] | 42.5 [38.9 to 46.4] | 6.0 [5.5 to 6.5] | 7.0 [6.1 to 8.0]
  A/TURK, Day 364 [N=151,147,100,NA] | 215.1 [190.3 to 243.3] | 35.4 [32.2 to 39.0] | 18.4 [16.3 to 20.9] | NA [NA to NA] — For D364, antibody titers were tabulated for GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group, GSK1562902A Formulation 1 - Havrix / Havrix Jr Group and GSK1562902A Formulation 2 - Havrix / Havrix Jr Group as required by the protocol.

5. Secondary Outcome: H5N1 HI Neutralizing Antibody Titres Against the A/Indonesia/5/2005 and A/Turkey/Turkey/01/2005 (H5N1 Virus) Strains
Description: Antibody titers were given as GMTs. A/Indonesia/5/2005 = A/INDO and A/Turkey/Turkey/01/2005 = A/TURK.
Time Frame: At Days 0, 42, 182, 192, 364
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group | GSK1562902A Formulation 1 - Havrix / Havrix Jr Group | GSK1562902A Formulation 2 - Havrix / Havrix Jr Group | Havrix / Havrix Jr Group
Number analyzed (Participants) | 151 | 147 | 100 | 102
Titer
  A/INDO, Day 0 [N=149,145,98,99] | 16.6 [15.4 to 17.9] | 16.0 [15.0 to 17.0] | 15.3 [14.4 to 16.3] | 16.0 [14.9 to 17.3]
  A/INDO,Day 42 [N=150,146,99,100] | 726.8 [646.1 to 817.6] | 804.1 [710.8 to 909.5] | 15.3 [14.4 to 16.4] | 17.0 [15.1 to 19.1]
  A/INDO, Day 182 [N=151,147,100,102] | 133.3 [125.2 to 142.0] | 140.7 [132.1 to 149.8] | 15.0 [14.2 to 15.8] | 14.7 [14.0 to 15.5]
  A/INDO, Day 192 [N=149,NA,99,NA] | 2128.0 [1864.0 to 2429.5] | NA [NA to NA] — For D192 , antibody titers were tabulated for GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group and GSK1562902A Formulation 2 - Havrix / Havrix Jr Group as required by the protocol. | 38.6 [33.7 to 44.1] | NA [NA to NA] — For D192 , antibody titers were tabulated for GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group and GSK1562902A Formulation 2 - Havrix / Havrix Jr Group as required by the protocol.
  A/INDO, Day 364 [N=149,147,100,NA] | 523.1 [452.9 to 604.2] | 132.7 [123.9 to 142.2] | 30.4 [26.8 to 34.4] | NA [NA to NA] — For D364, antibody titers were tabulated for GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group, GSK1562902A Formulation 1 - Havrix / Havrix Jr Group and GSK1562902A Formulation 2 - Havrix / Havrix Jr Group as required by the protocol.
  A/TURK, Day 0, [N=149,145,98,100] | 16.4 [15.3 to 17.6] | 15.9 [15.0 to 16.9] | 15.6 [14.5 to 16.8] | 17.3 [15.8 to 19.0]
  A/TURK, Day 42, [N=150,146,98,100] | 155.7 [141.9 to 171.0] | 162.7 [147.8 to 179.2] | 16.0 [14.7 to 17.5] | 17.6 [15.9 to 19.5]
  A/TURK, Day 182, [N=151,147,100,101] | 85.3 [79.7 to 91.2] | 85.1 [79.2 to 91.3] | 15.7 [14.6 to 16.8] | 15.5 [14.5 to 16.5]
  A/TURK, Day 192, [N=150,NA,100,NA] | 1420.4 [1229.6 to 1640.8] | NA [NA to NA] — For D192 , antibody titers were tabulated for GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group and GSK1562902A Formulation 2 - Havrix / Havrix Jr Group as required by the protocol. | 68.3 [58.2 to 80.2] | NA [NA to NA] — For D192 , antibody titers were tabulated for GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group and GSK1562902A Formulation 2 - Havrix / Havrix Jr Group as required by the protocol.
  A/TURK, Day 364, [N=149,145,98,NA] | 415.2 [359.2 to 479.9] | 99.9 [92.6 to 107.9] | 67.1 [59.6 to 75.5] | NA [NA to NA] — For D364, antibody titers were tabulated for GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group, GSK1562902A Formulation 1 - Havrix / Havrix Jr Group and GSK1562902A Formulation 2 - Havrix / Havrix Jr Group as required by the protocol.

6. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited Local Symptoms.
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site. Relationship analysis was not performed.
Time Frame: During a 7-day (Day 0-6) follow-up period after each vaccination
Population: The analysis was based on the Total vaccinated Cohort, which included all vaccinated subjects with at least 1 vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group | GSK1562902A Formulation 1 - Havrix / Havrix Jr Group | GSK1562902A Formulation 2 - Havrix / Havrix Jr Group | Havrix / Havrix Jr Group
Number analyzed (Participants) | 156 | 156 | 104 | 104
Subjects
  Any Pain, D1 [N=156,156,104,104] | 106 | 112 | 45 | 43
  Grade 3 Pain, D1 [N=156,156,104,104] | 2 | 3 | 1 | 1
  Any Redness, D1 [N=156,156,104,104] | 0 | 1 | 0 | 1
  Grade 3 Redness, D1 [N=156,156,104,104] | 0 | 0 | 0 | 0
  Any Swelling, D1 [N=156,156,104,104] | 9 | 9 | 0 | 1
  Grade 3 Swelling, D1 [N=156,156,104,104] | 0 | 0 | 0 | 0
  Any Pain, D2 [N=156,156,104,103] | 93 | 103 | 65 | 29
  Grade 3 Pain, D2 [N=156,156,104,103] | 3 | 0 | 0 | 0
  Any Redness, D2 [N=156,156,104,103] | 3 | 1 | 1 | 1
  Grade 3 Redness, D2 [N=156,156,104,103] | 0 | 0 | 0 | 0
  Any Swelling, D2 [N=156,156,104,103] | 7 | 7 | 2 | 1
  Grade 3 Swelling, D2 [N=156,156,104,103] | 0 | 0 | 0 | 0
  Any Pain, D3 [N=156,154,0,0] | 105 | 52 | 0 | 0
  Grade 3 Pain, D3 [N=156,154,0,0] | 0 | 0 | 0 | 0
  Any Redness, D3 [N=156,154,0,0] | 1 | 0 | 0 | 0
  Grade 3 Redness, D3 [N=156,154,0,0] | 0 | 0 | 0 | 0
  Any Swelling, D3 [N=156,154,0,0] | 4 | 0 | 0 | 0
  Grade 3 Swelling, D3 [N=156,1540,0] | 0 | 0 | 0 | 0
  Any Pain, Across [N=156,156,104,104] | 127 | 129 | 73 | 53
  Grade 3 Pain, Across [N=156,156,104,104] | 5 | 3 | 1 | 1
  Any Redness, Across [N=156,156,104,104] | 4 | 2 | 1 | 1
  Grade 3 Redness, Across [N=156,156,104,104] | 0 | 0 | 0 | 0
  Any Swelling, Across [N=156,156,104,104] | 15 | 13 | 2 | 1
  Grade 3 Swelling, Across [N=156,156,104,104] | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms.
Description: Assessed solicited general symptoms were diarrhea/vomiting, drowsiness, irritability/fussiness, loss of appetite and temperature [defined as axillary temperature equal to or above 38 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination. The symptoms were assessed for subjects aged less than 6 years.
Time Frame: During a 7-day (Day 0-6) follow-up period after each vaccination
Population: The analysis was based on subjects aged less than 6 years, comprised in the Total vaccinated Cohort, which included all vaccinated subjects with at least 1 vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group | GSK1562902A Formulation 1 - Havrix / Havrix Jr Group | GSK1562902A Formulation 2 - Havrix / Havrix Jr Group | Havrix / Havrix Jr Group
Number analyzed (Participants) | 30 | 31 | 22 | 24
Subjects
  Any diarrhoea/vomiting | 2 | 3 | 2 | 0
  Grade 3 diarrhoea/vomiting | 0 | 0 | 0 | 0
  Related diarrhoea/vomiting | 2 | 3 | 2 | 0
  Any drowsiness | 5 | 8 | 3 | 2
  Grade 3 drowsiness | 0 | 2 | 0 | 0
  Related drowsiness | 5 | 8 | 3 | 2
  Any irritability / fussiness | 8 | 10 | 3 | 1
  Grade 3 irritability / fussiness | 0 | 0 | 0 | 0
  Related irritability / fussiness | 8 | 10 | 3 | 1
  Any loss of appetite | 8 | 9 | 3 | 1
  Grade 3 loss of appetite | 0 | 0 | 0 | 0
  Related loss of appetite | 8 | 8 | 3 | 1
  Any temperature | 12 | 11 | 1 | 0
  Grade 3 temperature | 2 | 4 | 1 | 0
  Related temperature | 11 | 10 | 1 | 0

8. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms.
Description: Assessed solicited general symptoms were arthralgia, fatigue, gastrointestinal symptoms, headache, myalgia and temperature[defined as axillary temperature equal to or above 38 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination. The symptoms were assessed for subjects aged 6 years or more.
Time Frame: During a 7-day (Day 0-6) follow-up period after vaccination
Population: The analysis was based on subjects aged 6 years or more, comprised in the Total vaccinated Cohort, which included all vaccinated subjects with at least 1 vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group | GSK1562902A Formulation 1 - Havrix / Havrix Jr Group | GSK1562902A Formulation 2 - Havrix / Havrix Jr Group | Havrix / Havrix Jr Group
Number analyzed (Participants) | 126 | 125 | 82 | 80
Subjects
  Any Arthralgia, D1 [N=126,125,82,80] | 13 | 20 | 7 | 8
  Grade 3 Arthralgia, D1 [N=126,125,82,80] | 0 | 0 | 0 | 0
  Related Arthralgia, D1 [N=126,125,82,80] | 12 | 19 | 7 | 7
  Any Fatigue, D1 [N=126,125,82,80] | 16 | 16 | 8 | 8
  Grade 3 Fatigue, D1 [N=126,125,82,80] | 0 | 0 | 0 | 0
  Related Fatigue, D1 [N=126,125,82,80] | 15 | 16 | 8 | 7
  Any Gastrointestinal symptoms,D1 [N=126,125,82,80] | 9 | 5 | 6 | 7
  Grade 3 Gastrointestinal ,D1 [N=126,125,82,80] | 0 | 0 | 0 | 1
  Related Gastrointestinal ,D1 [N=126,125,82,80] | 7 | 5 | 6 | 6
  Any Headache, D1 [N=126,125,82,80] | 31 | 24 | 14 | 19
  Grade 3 Headache, D1 [N=126,125,82,80] | 1 | 1 | 0 | 0
  Related Headache, D1 [N=126,125,82,80] | 30 | 23 | 12 | 17
  Any Myalgia, D1 [N=126,125,82,80] | 14 | 23 | 8 | 11
  Grade 3 Myalgia, D1 [N=126,125,82,80] | 0 | 0 | 0 | 0
  Related Myalgia, D1 [N=126,125,82,80] | 14 | 22 | 8 | 10
  Any Temperature/(Axillary), D1 [N=126,125,82,80] | 10 | 2 | 6 | 7
  Grade 3 Temperature/(Axillary),D1[N=126,125,82,80] | 1 | 1 | 2 | 1
  Related Temperature/(Axillary),D1[N=126,125,82,80] | 8 | 1 | 3 | 5
  Any Arthralgia, D2 [N=126,125,82,79] | 11 | 18 | 5 | 3
  Grade 3 Arthralgia, D2 [N=126,125,82,79] | 0 | 0 | 0 | 0
  Related Arthralgia, D2 [N=126,125,82,79] | 11 | 18 | 5 | 3
  Any Fatigue, D2 [N=126,125,82,79] | 12 | 7 | 5 | 3
  Grade 3 Fatigue, D2 [N=126,125,82,79] | 0 | 0 | 0 | 0
  Related Fatigue, D2 [N=126,125,82,79] | 12 | 7 | 5 | 3
  Any Gastrointestinal symptoms, D2[N=126,125,82,79] | 6 | 7 | 3 | 1
  Grade 3 Gastrointestinal, D2 [N=126,125,82,79] | 0 | 0 | 0 | 0
  Related Gastrointestinal, D2 [N=126,125,82,79] | 6 | 7 | 3 | 1
  Any Headache, D2 [N=126,125,82,79] | 40 | 37 | 8 | 12
  Grade 3 Headache, D2 [N=126,125,82,79] | 4 | 0 | 0 | 1
  Related Headache, D2 [N=126,125,82,79] | 39 | 37 | 8 | 12
  Any Myalgia, D2 [N=126,125,82,79] | 13 | 20 | 7 | 3
  Grade 3 Myalgia, D2 [N=126,125,82,79] | 0 | 0 | 0 | 0
  Related Myalgia, D2 [N=126,125,82,79] | 13 | 19 | 7 | 3
  Any Temperature (Axillary), D2 [N=126,125,82,79] | 11 | 17 | 4 | 0
  Grade 3 Temperature(Axillary),D2 [N=126,125,82,79] | 2 | 5 | 0 | 0
  Related Temperature(Axillary),D2 [N=126,125,82,79] | 10 | 15 | 4 | 0
  Any Arthralgia, D3 [N=126,124,0,0] | 19 | 3 | 0 | 0
  Grade 3 Arthralgia, D3 [N=126,124,0,0] | 0 | 0 | 0 | 0
  Related Arthralgia, D3 [N=126,124,0,0] | 19 | 3 | 0 | 0
  Any Fatigue, D3 [N=126,124,0,0] | 15 | 8 | 0 | 0
  Grade 3 Fatigue, D3 [N=126,124,0,0] | 0 | 0 | 0 | 0
  Related Fatigue, D3 [N=126,124,0,0] | 15 | 8 | 0 | 0
  Any Gastrointestinal, D3 [N=126,124,0,0] | 4 | 6 | 0 | 0
  Grade 3 Gastrointestinal, D3 [N=126,124,0,0] | 0 | 0 | 0 | 0
  Related Gastrointestinal, D3 [N=126,124,0,0] | 4 | 6 | 0 | 0
  Any Headache, D3 [N=126,124,0,0] | 39 | 17 | 0 | 0
  Grade 3 Headache, D3 [N=126,124,0,0] | 1 | 0 | 0 | 0
  Related Headache Headache, D3 [N=126,124,0,0] | 39 | 17 | 0 | 0
  Any Myalgia, D3 [N=126,124,0,0] | 15 | 2 | 0 | 0
  Grade 3 Myalgia, D3 [N=126,124,0,0] | 0 | 0 | 0 | 0
  Related Myalgia, D3 [N=126,124,0,0] | 15 | 2 | 0 | 0
  Any Temperature (Axillary), D3 [N=126,124,0,0] | 7 | 2 | 0 | 0
  Grade 3 Temperature (Axillary), D3 [N=126,124,0,0] | 0 | 0 | 0 | 0
  Related Temperature (Axillary), D3 [N=126,124,0,0] | 7 | 2 | 0 | 0
  Any Arthralgia, Across [N=126,125,82,80] | 33 | 31 | 11 | 11
  Grade 3 Arthralgia, Across [N=126,125,82,80] | 0 | 0 | 0 | 0
  Related Arthralgia, Across [N=126,125,82,80] | 32 | 30 | 11 | 10
  Any Fatigue, Across [N=126,125,82,80] | 28 | 22 | 10 | 10
  Grade 3 Fatigue, Across [N=126,125,82,80] | 0 | 0 | 0 | 0
  Related Fatigue, Across [N=126,125,82,80] | 28 | 22 | 10 | 9
  Any Gastrointestinal, Across [N=126,125,82,80] | 16 | 12 | 8 | 7
  Grade 3 Gastrointestinal, Across [N=126,125,82,80] | 0 | 0 | 0 | 1
  Related Gastrointestinal, Across [N=126,125,82,80] | 15 | 12 | 8 | 6
  Any Headache, Across [N=126,125,82,80] | 63 | 52 | 20 | 24
  Grade 3 Headache, Across [N=126,125,82,80] | 5 | 1 | 0 | 1
  Related Headache, Across [N=126,125,82,80] | 62 | 51 | 18 | 22
  Any Myalgia, Across [N=126,125,82,80] | 29 | 33 | 13 | 13
  Grade 3 Myalgia, Across [N=126,125,82,80] | 0 | 0 | 0 | 0
  Related Myalgia, Across [N=126,125,82,80] | 29 | 31 | 13 | 12
  Any Temperature/(Axillary),Across[N=126,125,82,80] | 23 | 19 | 10 | 7
  Grade 3 Temperature, Across [N=126,125,82,80] | 3 | 6 | 2 | 1
  Related Temperature, Across [N=126,125,82,80] | 20 | 16 | 7 | 5

9. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs).
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During a 21-day (Days 0 - 20) follow-up period after vaccination
Population: as for outcome 6
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group | GSK1562902A Formulation 1 - Havrix / Havrix Jr Group | GSK1562902A Formulation 2 - Havrix / Havrix Jr Group | Havrix / Havrix Jr Group
Number analyzed (Participants) | 156 | 156 | 104 | 104
Subjects
  Any AEs | 60 | 82 | 35 | 20
  Grade 3 AEs | 1 | 1 | NA — Grade 3 AEs were not reported in this group. | NA — Grade 3 AEs were not reported in this group.
  Related AEs | 12 | 7 | 7 | 3

10. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs).
Description: as for outcome 9
Time Frame: During Day 0 to Telephone Contact (TC) Day 84 overall.
Population: as for outcome 6
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group | GSK1562902A Formulation 1 - Havrix / Havrix Jr Group | GSK1562902A Formulation 2 - Havrix / Havrix Jr Group | Havrix / Havrix Jr Group
Number analyzed (Participants) | 156 | 156 | 104 | 104
Subjects
  Any AEs | 75 | 92 | 59 | 50
  Grade 3 AEs | 2 | 0 | 1 | 1
  Related AEs | 7 | 6 | 3 | 3

11. Secondary Outcome: Number of Subjects With Any Potential Immune-Mediated Diseases (pIMDs)
Time Frame: During the entire study period (Day 0 to 364)
Population: as for outcome 6
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group | GSK1562902A Formulation 1 - Havrix / Havrix Jr Group | GSK1562902A Formulation 2 - Havrix / Havrix Jr Group | Havrix / Havrix Jr Group
Number analyzed (Participants) | 156 | 156 | 104 | 104
Subjects | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs).
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (Day 0 to 364)
Population: as for outcome 6
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group | GSK1562902A Formulation 1 - Havrix / Havrix Jr Group | GSK1562902A Formulation 2 - Havrix / Havrix Jr Group | Havrix / Havrix Jr Group
Number analyzed (Participants) | 156 | 156 | 104 | 104
Subjects | 4 | 1 | 0 | 0

13. Secondary Outcome: Number of Subjects With Anti-H5N1 Antibodies Above the Cut Off Values ≥1:10
Description: Seropositivity rates against the A/Indonesia/5/2005 (H5N1 virus) strain, were tabulated on Days 0,42,182 for all subjects, 192 for GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group, GSK1562902A Formulation 2 - Havrix / Havrix Jr Group and 364 for GSK1562902A Formulation 1 - Havrix / Havrix Jr Group and GSK1562902A Formulation 1 - Havrix / Havrix Jr Group.
  Seropositivity rates against the A/turkey/Turkey/01/2005 (H5N1 virus) strain, were tabulated on Days 182, 192 and 364.
Time Frame: At Days 0, 42, 182, 192 and 364
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group | GSK1562902A Formulation 1 - Havrix / Havrix Jr Group | GSK1562902A Formulation 2 - Havrix / Havrix Jr Group | Havrix / Havrix Jr Group
Number analyzed (Participants) | 155 | 152 | 103 | 101
Subjects
  A/INDO, Day 0 [N=155,152,103,101] | 22 | 15 | 8 | 14
  A/INDO, Day 42 [N=155,152,103,101] | 155 | 151 | 9 | 19
  A/INDO, Day 182 [N=155,152,103,101] | 154 | 152 | 2 | 12
  A/INDO, Day 192 [N=127,0,84,0] | 127 | 0 | 37 | 0
  A/INDO, Day 364 [N=151,147,100,0] | 151 | 147 | 57 | 0
  A/TURK, Day 182 [N=127,152,84,101] | 126 | 152 | 17 | 26
  A/TURK, Day 364 [N=151,147,100,0] | 151 | 147 | 95 | 0

14. Secondary Outcome: Number of Seroconverted Subjects Against the A/Indonesia/05/2005 Strains of H5N1 Influenza Disease
Description: A seroconverted subject was defined as a vaccinee with either a pre-vaccination titer less than (<) 1:10 and a post-vaccination titer ≥ 1:40, or a pre-vaccination titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer.
  Seroconversion rates against the A/Indonesia/05/2005 (H5N1 VIRUS) strain were tabulated on Days 0,42,182 for all subjects, 192 for GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group, GSK1562902A Formulation 2 - Havrix / Havrix Jr Group and 364 for GSK1562902A Formulation 1 - Havrix / Havrix Jr Group and GSK1562902A Formulation 1 - Havrix / Havrix Jr Group.
Time Frame: At Days 42, 182, 192 and 364
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group | GSK1562902A Formulation 1 - Havrix / Havrix Jr Group | GSK1562902A Formulation 2 - Havrix / Havrix Jr Group | Havrix / Havrix Jr Group
Number analyzed (Participants) | 155 | 152 | 103 | 101
Subjects
  A/INDO, Day 42 [N=155,152,103,101] | 154 | 151 | 1 | 1
  A/INDO, Day 182 [N=155,152,103,101] | 122 | 121 | 0 | 0
  A/INDO, Day 192 [N=127,0,84,0] | 127 | 0 | 3 | 0
  A/INDO, Day 364 [N=151,147,100,0] | 151 | 100 | 1 | 0

15. Secondary Outcome: Number of Seroprotected Subjects Against the A/Indonesia/05/2005 and A/Turkey/Turkey/01/2005 Strains of H5N1 Influenza Disease
Description: A seroprotected subject was defined as a subject with a serum HI titer greater than or equal to 1:40 that usually is accepted as indicating protection.
  Seroprotection rates against the A/Indonesia/5/2005 (H5N1 virus) strain, were tabulated 95% CI on Days 0,42,182 for all subjects, 192 for GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group, GSK1562902A Formulation 2 -Havrix / Havrix Jr Group and 364 for GSK1562902A Formulation 1 - Havrix / Havrix Jr Group and GSK1562902A Formulation 1 - Havrix / Havrix Jr Group.
  Seroprotection rates against the A/turkey/Turkey/01/2005 (H5N1 virus) strain, were tabulated on Days 182 and 192.
Time Frame: At Days 0,42, 182, 192 and 364
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group | GSK1562902A Formulation 1 - Havrix / Havrix Jr Group | GSK1562902A Formulation 2 - Havrix / Havrix Jr Group | Havrix / Havrix Jr Group
Number analyzed (Participants) | 155 | 152 | 103 | 101
Subjects
  A/INDO, Day 0 [N=155,152,103,101] | 0 | 0 | 2 | 1
  A/INDO, Day 42 [N=155,152,103,101] | 154 | 151 | 2 | 1
  A/INDO, Day 182 [N=155,152,103,101] | 125 | 122 | 0 | 0
  A/INDO, Day 192 [N=127,0,84,0] | 127 | 0 | 3 | 0
  A/INDO, Day 364 [N=151,147,100,0] | 151 | 102 | 1 | 0
  A/TURK, Day 182 [N=127,0,84,0] | 73 | 0 | 1 | 0
  A/TURK, Day 192 [N=127,0,84,0] | 127 | 0 | 28 | 0

16. Secondary Outcome: Mean Geometric Increase for Anti-H5N1 Antibody Titers
Description: MGI against the A/Indonesia/05/2005 (H5N1 VIRUS) strain were tabulated on Days 0,42,182 for all subjects, 192 for GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group, GSK1562902A Formulation 2 - Havrix / Havrix Jr Group and 364 for GSK1562902A Formulation 1 - Havrix / Havrix Jr Group and GSK1562902A Formulation 1 - Havrix / Havrix Jr Group.
  MGI against the A/turkey/Turkey/01/2005 (H5N1 virus) strain were tabulated on Days 42, 182 and 364.
Time Frame: At Days 42, 182, 192 and 364
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group | GSK1562902A Formulation 1 - Havrix / Havrix Jr Group | GSK1562902A Formulation 2 - Havrix / Havrix Jr Group | Havrix / Havrix Jr Group
Number analyzed (Participants) | 155 | 152 | 103 | 101
Titer
  A/INDO, Day 42 [N=155,152,103,101] | 96.9 [84.9 to 110.4] | 108.4 [94.2 to 124.7] | 1 [1 to 1.1] | 1.1 [0.9 to 1.2]
  A/INDO, Day 182 [N=155,152,103,101] | 9.1 [8.3 to 10.1] | 9.8 [9 to 10.8] | 0.9 [0.9 to 1] | 1 [0.9 to 1.1]
  A/INDO, Day 192 [N=127,0,84,0] | 117.7 [103 to 134.5] | NA [NA to NA] — MGI against the A/Indonesia/05/2005 (H5N1 VIRUS) strain were tabulated on Day 192 for GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group and GSK1562902A Formulation 2 - Havrix / Havrix Jr Group only. | 1.4 [1.2 to 1.6] | NA [NA to NA] — MGI against the A/Indonesia/05/2005 (H5N1 VIRUS) strain were tabulated on Day 192 for GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group and GSK1562902A Formulation 2 - Havrix / Havrix Jr Group only.
  A/INDO, Day 364 [N=151,147,100,0] | 36.2 [32 to 40.9] | 7.4 [6.7 to 8.2] | 1.6 [1.4 to 1.7] | NA [NA to NA] — MGI against the A/Indonesia/05/2005 (H5N1 VIRUS) strain were tabulated on Day 364 for GSK1562902A Formulation 1 and 2-Havrix/Havrix Jr Group, GSK1562902A Formulation 1-Havrix/Havrix Jr Group and GSK1562902A Formulation 2-Havrix/Havrix Jr Group only.
  A/TURK, Day 42 [N=155,152,103,101] | 27.7 [24 to 31.9] | 33.1 [28.6 to 38.3] | 1.1 [1 to 1.3] | 1.2 [1.1 to 1.3]
  A/TURK, Day 182 [N=155,152,103,101] | 5.6 [5 to 6.3] | 6.6 [6 to 7.4] | 1 [0.9 to 1.1] | 1 [0.9 to 1.1]
  A/TURK, Day 364 [N=151,147,100,0] | 31.4 [26.9 to 36.7] | 5.6 [5 to 6.3] | 3 [2.6 to 3.4] | NA [NA to NA] — MGI against the A/turkey/Turkey/01/2005 (H5N1) strain were tabulated on Day 364 for GSK1562902A Formulation 1 and 2-Havrix/Havrix Jr Group, GSK1562902A Formulation 1-Havrix/Havrix Jr Group and GSK1562902A Formulation 2-Havrix/Havrix Jr Group only

17. Secondary Outcome: Number of Seroconverted Subjects Against the A/Turkey/Turkey/01/2005 Strains of H5N1 Influenza Disease
Description: Booster seroconversion rates against the A/turkey/Turkey/01/2005 (H5N1 VIRUS) strain were tabulated on Days 192 and 364.
  This outcome concerns solely subjects in the GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group and GSK1562902A Formulation 2 - Havrix / Havrix Jr Group as required by the protocol.
Time Frame: At Days 192 and 364
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group | GSK1562902A Formulation 2 - Havrix / Havrix Jr Group
Number analyzed (Participants) | 151 | 100
Subjects
  A/TURK, Day 192 [N=127,84] | 127 | 27
  A/TURK, Day 364 [N=151,100] | 105 | 18

18. Secondary Outcome: Booster Factor for Hemagglutination Inhibition (HI) Antibodies Against the A/Turkey/Turkey/01/2005 Strain of H5N1 Influenza Disease
Description: Boooster factor against the A/turkey/Turkey/01/2005 (H5N1 VIRUS) strain were tabulated 95% CI on Days 192,364. This outcome concerns solely subjects in the GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group and GSK1562902A Formulation 2 - Havrix / Havrix Jr Group as required by the protocol.
Time Frame: At Days 192 and 364
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group | GSK1562902A Formulation 2 - Havrix / Havrix Jr Group
Number analyzed (Participants) | 151 | 100
Titer
  A/TURK, Day 192 [N=127,84] | 18.6 [16.3 to 21.3] | 4.1 [3.3 to 5.2]
  A/TURK, Day 364 [N=151,100] | 5.6 [5 to 6.3] | 3 [2.7 to 3.4]

19. Secondary Outcome: Number of Subjects With Neutralizing Anti-H5N1 Antibody Titers
Description: Seropositivity rates against the A/Indonesia/5/2005 (H5N1 virus) strain, were tabulated on Days 0,42,182 for all subjects, 192 for GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group, GSK1562902A Formulation 2 - Havrix / Havrix Jr Group and 364 for GSK1562902A Formulation 1 - Havrix / Havrix Jr Group and GSK1562902A Formulation 1 - Havrix / Havrix Jr Group.
  Seropositivity rates against the A/turkey/Turkey/01/2005 (H5N1 virus) strain, were tabulated on Days 0, 42,182, 192 and 364.
Time Frame: At Days 0, 42, 182 192 and 364
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group | GSK1562902A Formulation 1 - Havrix / Havrix Jr Group | GSK1562902A Formulation 2 - Havrix / Havrix Jr Group | Havrix / Havrix Jr Group
Number analyzed (Participants) | 151 | 147 | 100 | 102
Subjects
  A/INDO, Day 0 [N=149,145,98,99] | 22 | 17 | 8 | 14
  A/INDO,Day 42 [N=150,146,99,100] | 150 | 146 | 9 | 15
  A/INDO, Day 182 [N=151,147,100,102] | 150 | 147 | 7 | 4
  A/INDO, Day 192 [N=149,0,99,0] | 149 | 0 | 75 | 0
  A/INDO, Day 364 [N=149,147,100,0] | 149 | 147 | 73 | 0
  A/TURK, Day 0, [N=149,145,98,100] | 21 | 18 | 8 | 19
  A/TURK, Day 42, [N=150,146,98,100] | 150 | 145 | 10 | 20
  A/TURK, Day 182, [N=151,147,100,101] | 150 | 145 | 11 | 10
  A/TURK, Day 192, [N=150,0,100,0] | 150 | 0 | 90 | 0
  A/TURK, Day 364, [N=149,145,98,0] | 149 | 145 | 95 | 0

20. Secondary Outcome: Number of Subjects With Vaccine Response Rates (VRR) for H5N1 Neutralizing Antibodies
Time Frame: At Days 42, 182 192 and 364
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group | GSK1562902A Formulation 1 - Havrix / Havrix Jr Group | GSK1562902A Formulation 2 - Havrix / Havrix Jr Group | Havrix / Havrix Jr Group
Number analyzed (Participants) | 149 | 145 | 98 | 98
Subjects
  A/INDO,Day 42 [N=149,144,98,98] | 147 | 142 | 0 | 2
  A/INDO, Day 182 [N=149,145,98,98] | 127 | 115 | 0 | 0
  A/INDO, Day 192 [N=147,0,97,0] | 147 | 0 | 5 | 0
  A/INDO, Day 364 [N=148,145,98,0] | 144 | 126 | 8 | 0

21. Secondary Outcome: Number of Subjects With Booster Vaccine Response for H5N1 Neutralizing Antibodies
Description: This outcome concerns solely subjects in the GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group and GSK1562902A Formulation 2 - Havrix / Havrix Jr Group as required by the protocol.
Time Frame: At Days 192 and 364
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group | GSK1562902A Formulation 2 - Havrix / Havrix Jr Group
Number analyzed (Participants) | 150 | 100
Subjects
  A/TURK, Day 192, [N=150,100] | 141 | 38
  A/TURK, Day 364, [N=149,98] | 86 | 36

ADVERSE EVENTS:
Time Frame: Systematically-assessed symptoms: during the 7 days after each vaccination; unsolicited AEs: within 21 days after each vaccination and from Day 0 to Day 84. SAEs were collected throughout the study from Day 0 to Day 364.
Description: Solicited general symptoms were assessed in subjects aged less than 6 years and in subjects aged 6 years and more as required by the protocol.
Arm/Group | GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group | GSK1562902A Formulation 1 - Havrix / Havrix Jr Group | GSK1562902A Formulation 2 - Havrix / Havrix Jr Group | Havrix / Havrix Jr Group
Serious Adverse Events (participants affected / at risk) | 4/156 | 1/156 | 0/104 | 0/104
Other Adverse Events (participants affected / at risk) | 138/156 | 145/156 | 87/104 | 77/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group (N=156) | GSK1562902A Formulation 1 - Havrix / Havrix Jr Group (N=156) | GSK1562902A Formulation 2 - Havrix / Havrix Jr Group (N=104) | Havrix / Havrix Jr Group (N=104)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Open wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Typhoid fever (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | GSK1562902A Formulation 1 and 2 - Havrix / Havrix Jr Group (N=156) | GSK1562902A Formulation 1 - Havrix / Havrix Jr Group (N=156) | GSK1562902A Formulation 2 - Havrix / Havrix Jr Group (N=104) | Havrix / Havrix Jr Group (N=104)
Pain (General disorders) | 127 | 129 | 73 | 53
Swelling (General disorders) | 15 | 13 | 2 | 1
Diarrhoea/vomiting (General disorders) | 2/30 | 3/31 | 2/22 | 0/24 — AE reported for subjects aged less than 6 years.
Drowsiness (General disorders) | 5/30 | 8/31 | 3/22 | 2/24 — AE reported for subjects aged less than 6 years.
Irritability / fussiness (General disorders) | 8/30 | 10/31 | 3/22 | 1/24 — AE reported for subjects aged less than 6 years.
Loss of appetite (General disorders) | 8/30 | 9/31 | 3/22 | 1/24 — AE reported for subjects aged less than 6 years.
Temperature (General disorders) | 12/30 | 11/31 | 1/22 | 0/24 — AE reported for subjects aged less than 6 years.
Arthralgia (General disorders) | 33/126 | 31/125 | 11/82 | 11/80 — AE reported for subjects aged 6 years or more.
Fatigue (General disorders) | 28/126 | 22/125 | 10/82 | 10/80 — AE reported for subjects aged 6 years or more.
Gastrointestinal symptoms (General disorders) | 16/126 | 12/125 | 8/82 | 7/80 — AE reported for subjects aged 6 years or more.
Headache (General disorders) | 63/126 | 52/125 | 20/82 | 24/80 — AE reported for subjects aged 6 years or more.
Myalgia (General disorders) | 29/126 | 33/125 | 13/82 | 13/80 — AE reported for subjects aged 6 years or more.
Temperature (General disorders) | 23/126 | 19/125 | 10/82 | 7/80 — AE reported for subjects aged 6 years or more.
Upper respiratory tract infection (Infections and infestations) | 31 | 54 | 9 | 9 — AE reported within 21 days post-vaccination.
Viral infection (Infections and infestations) | 2 | 10 | 7 | 2 — AE reported within 21 days post-vaccination.
Rhinitis (Infections and infestations) | 5 | 5 | 6 | 2 — AE reported within 21 days post-vaccination.
Upper respiratory tract infection (Infections and infestations) | 45 | 63 | 31 | 27 — AE reported from Day 0 up to Day 84 post-vaccination.
Nasopharyngitis (Infections and infestations) | 3 | 8 | 3 | 6 — AE reported from Day 0 up to Day 84 post-vaccination.
Viral infection (Infections and infestations) | 10 | 20 | 18 | 10 — AE reported from Day 0 up to Day 84 post-vaccination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.